CLINICAL TRIAL: NCT00317889
Title: Compaction THA Bilateral
Brief Title: Compaction Total Hip Arthroplasty (THA) Bilateral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON-04-002b-SKO
Record Dates: First submitted 2006-04-23; First posted 2006-04-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Coxarthrosis
Keywords: THA
MeSH Terms: conditions — Osteoarthritis, Hip

ARMS (2):
- Compaction (Experimental): Compaction technique for femoral bone preparation prior to cementless femoral stem insertion.
  Interventions: Procedure: Bone preparation technique: compaction
- Broaching (Active Comparator): Broaching technique for femoral bone preparation prior to cementless femoral stem insertion.
  Interventions: Procedure: Bone preparation technique: broaching

INTERVENTIONS:
Procedure: Bone preparation technique: compaction
  Other Names: No other names.
  Arms: Compaction
Procedure: Bone preparation technique: broaching
  Other Names: No other names.
  Arms: Broaching

SUMMARY:
This is a prospective, randomized study comparing two different bone preparation techniques for insertion of a porous coated titanium cementless femoral stem. Patients receiving a bilateral total hip replacement are randomized to conventional broaching on one side and compaction on the other side.

Hypothesis: Compaction results in significantly less stem migration [evaluated by radiostereometric analysis (RSA)], less peri-prosthetic bone mineral density (BMD) loss [evaluated by dual energy x-ray absorptiometry (DEXA)], and a higher Harris hip score after two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary arthritis in the hip
* Patients with sufficient bone density to allow uncemented implantation of a femoral component
* Informed patient consent in writing

Exclusion Criteria:

* Patients with neuromuscular or vascular disease in the affected leg
* Patients found upon operation to be unsuited for uncemented acetabulum component
* Patients who regularly take non-steroidal anti-inflammatory drugs (NSAIDs) and cannot interrupt intake for the postoperative phase of the study
* Patients with fracture sequelae
* Female patients of childbearing capacity
* Hip joint dysplasia
* Sequelae to previous hip joint disorder in childhood.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Radiostereometric analysis | 5 and 10 years follow-up
  Stem subsidence (change) at 5 and 10 years measured with radiostereometric analysis

SECONDARY OUTCOMES:
Periprosthetic bone mineral density | 5 years follow-up
  Periprosthetic bone mineral density measured with Dual Energy X-ray Absorptiometry (DXA)

OTHER OUTCOMES:
Questionnaire | 5 years follow-up
  Questionnaire of hip function

CONTACTS AND LOCATIONS:
Overall Officials: Søren Kold, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Aalborg and Farsø, Aalborg, Denmark